CLINICAL TRIAL: NCT00853762
Title: An Open-label, Multicenter Phase II Extension of Study 28063 (ATAMS) to Obtain Long-term Follow-up Data in Subjects With Relapsing Multiple Sclerosis Treated With Atacicept for up to 5 Years (ATAMS-Extension)
Brief Title: Atacicept in Multiple Sclerosis Extension Study, Phase II
Acronym: ATAMS ext
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: EMD Serono voluntarily decided to terminate this trial after observing increased MS disease activity in trial 28063 ATAMS [Please refer to ATAMS]
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28851
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Atacicept 25 mg (With Loading) (Experimental)
  Interventions: Drug: Atacicept 25 mg
- Atacicept 75 mg (With Loading) (Experimental)
  Interventions: Drug: Atacicept 75 mg
- Atacicept 150 mg (With Loading) (Experimental)
  Interventions: Drug: Atacicept 150 mg
- Atacicept 150 mg (Without Loading) (Experimental)
  Interventions: Drug: Atacicept 150 mg

INTERVENTIONS:
Drug: Atacicept 25 mg — Subjects who received atacicept 25 milligram (mg) subcutaneously (SC) as loading dose twice weekly for first 4 weeks, followed by atacicept 25 mg SC for 32 weeks, in 28063 study will continue with atacicept 25 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
  Arms: Atacicept 25 mg (With Loading)
Drug: Atacicept 75 mg — Subjects who received atacicept 75 mg SC as loading dose twice weekly for first 4 weeks, followed by atacicept 75 mg SC for 32 weeks, in 28063 study will continued with atacicept 75 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
  Arms: Atacicept 75 mg (With Loading)
Drug: Atacicept 150 mg — Subjects who received atacicept 150 mg SC as loading dose twice weekly for first 4 weeks, followed by atacicept 150 mg SC for 32 weeks, in 28063 study will continue with atacicept 150 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
  Arms: Atacicept 150 mg (With Loading)
Drug: Atacicept 150 mg — Subjects who received placebo SC twice weekly for first 4 weeks, followed by placebo SC for 32 weeks, in 28063 study will continue with atacicept 150 mg (without loading dose) SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
  Arms: Atacicept 150 mg (Without Loading)

SUMMARY:
This study (28851) is a long-term follow-up study of subjects enrolled in ATAMS study 28063 (NCT00642902). The aim of this study is to monitor the safety and tolerability of atacicept administered for up to 5 years to subjects with relapsing multiple sclerosis (RMS).

This extension study consists of two parts. Part A will be double blind and Part B will be open label. During Part A, subjects initially randomized to atacicept will continue to receive the atacicept dose to which they have been randomized in study 28063 (ATAMS) once a week subcutaneously (under the skin). Subjects randomized to placebo in ATAMS will receive atacicept at 150 mg once a week subcutaneously during Part A. Once the results of ATAMS are available and the atacicept dose with the best benefit / risk ratio has been identified, all subjects will be switched to this dose and will continue the extension study open-label (Part B). Throughout the study, subjects and investigators will remain blinded with respect to initial and part A treatment allocation/dose.

ELIGIBILITY:
Inclusion Criteria:

* Participation in study 28063.
* Completion of Week 36 visit of the core study 28063.
* Willingness and ability to comply with study procedures for the duration of the study.
* Voluntary provision of written informed consent (including, for the USA, subject authorization under the Health Insurance Portability and Accountability Act (HIPAA)), given before any study-related procedure that is not part of normal medical care and with the understanding that the subject may withdraw consent at any time without prejudice to his or her future medical care.

Exclusion Criteria:

* Premature discontinuation of core study 28063.
* Subjects who meet criteria listed below will receive IMP in study 28851:

  * Subjects who are eligible for participation in extension study 28851 but do not meet these criteria will not be treated with IMP but will undergo scheduled visits, irrespective of their treatment.
* All subjects must satisfy the following criteria before Extension Study Day 1 (D1-EXT; defined as the first day of dosing in the extension study) to be eligible for treatment with IMP:

  * Eligibility for participation in extension study 28851.
  * For women of childbearing potential, a negative urine pregnancy test at eligibility assessment.
  * Female subjects of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for four (4) weeks before the first dose administered within the extension study, during the study and for twelve (12) weeks after the last dose of trial medication. Adequate contraception is defined as two barrier methods, or one barrier method with spermicide, or an intrauterine device, or use of a combined oral female hormonal contraceptive (or the definitions requested by health authorities and locally amended in the core study 28063). For the purposes of this trial, women of childbearing potential are defined as: "All female subjects after puberty unless they are post-menopausal for at least two years or are surgically sterile" (For Germany Only: Female subjects of childbearing potential must be willing to avoid pregnancy by using highly effective methods of contraception for approximately four (4) weeks prior to D1-EXT, during and for twelve (12) weeks after the last dose of trial medication. This requirement does not apply to surgically sterile subjects or to subjects who are postmenopausal for at least 2 years. Highly effective contraception is defined as any method or combination of methods which result in a low failure rate (i.e. less than (<) 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, sexual abstinence, vasectomized partner, 2 barrier methods, or 1 barrier method with spermicide)
* Willingness and ability to comply with study procedures for the duration of the study.
* To be eligible for treatment with investigational medicinal product (IMP) in study 28851, the subjects must not meet any of the following criteria:
* Non-eligibility for participation in extension study 28851 (premature discontinuation of core study 28063).
* Major protocol violation or non-compliance in the core study.
* Use of prohibited immunomodulatory / immunosuppressive therapies
* Serum immunoglobulin G (IgG) level <3 gram per liter (g/L) if the subject received atacicept in the core study, or serum IgG level <6 g/L if the subject received placebo in the core study (to protect the blinding of the core study, the IgG level will be communicated to the treating physician only if it is too low for extension study participation and only after all Week 36 assessments performed within the core study have been completed).
* Any condition, including laboratory findings that, in the opinion of the Investigator, constitutes a risk or a contraindication for participation in the extension study, or that could interfere with the study objectives, conduct or evaluation.
* Known active clinically significant acute or chronic infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives.
* Investigator judgement that treatment of the subject with atacicept in the extension study is not appropriate.
* Aspartate aminotransferase (AST), or alanine aminotransferase (ALT), or alkaline phosphatase (AP) level greater than (>)2.5 x upper limit of normal (ULN), or total bilirubin >1.5 x ULN at eligibility assessment.
* Clinically significant abnormality in any hematological test (e.g. hemoglobin <100 g/L (6.21 millimoles per liter [mmol/L]), white blood cells <3 x 10^9 per liter (/L), platelets <100 x 10^9/L) at eligibility assessment.
* Clinically significant abnormality on electrocardiogram (ECG) performed at eligibility assessment.
* Presence of uncontrolled or New York Health Association (NYHA) class 3 or 4 congestive heart failure at Week 36 of the core study.
* Moderate to severe renal impairment (creatinine clearance <50 milliliter per minute (mL/min) according to Cockcroft-Gault equation).
* Allergy or hypersensitivity to gadolinium (Gd).
* Allergy or hypersensitivity to atacicept or to any of the components of the formulated atacicept.
* Diagnosis or family history of Creutzfeldt-Jakob disease (CJD).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mikol, MD, PhD, Study Director — EMD Serono
Locations (47):
- United States (6):
  - Research Site, Phoenix, Arizona
  - Research Site, Northbrook, Illinois
  - Research Site, East Lansing, Michigan
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Australia (4):
  - Research Site, Box Hill VIC
  - Research Site, Fitzroy
  - Research Site, New Lambton
  - Research Site, Woodville
- Belgium (2):
  - Research Site, Diepenbeek
  - Research Site, Sijsele
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
- Czechia (2):
  - Research Site, Brno
  - Research Site, Hradec Králové
- France (2):
  - Research Site, Caen
  - Research Site, Saint-Herblain
- Germany (2):
  - Research Site, Bochum
  - Research Site, Düsseldorf
- Research Site, Beirut, Lebanon
- Research Site, Kaunas, Lithuania
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
- Research Site, Winston Salem, New Caledonia
- Russia (7):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Vladimir
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Stockholm, Sweden
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Innsbruck
  - Research Site, Zurich
- Ukraine (4):
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Uzhhorod
- United Kingdom (3):
  - Research Site, London
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Kappos L, Hartung HP, Freedman MS, Boyko A, Radu EW, Mikol DD, Lamarine M, Hyvert Y, Freudensprung U, Plitz T, van Beek J; ATAMS Study Group. Atacicept in multiple sclerosis (ATAMS): a randomised, placebo-controlled, double-blind, phase 2 trial. Lancet Neurol. 2014 Apr;13(4):353-63. doi: 10.1016/S1474-4422(14)70028-6. Epub 2014 Mar 6. PMID 24613349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): 03 March 2009/13 August 2009. Last participant completed: 09 September 2009.
Pre-assignment Details: A total of 324 subjects were screened and 255 were enrolled in ATAMS (28063; NCT00642902). Overall, 75 subjects randomized and treated in ATAMS were eligible to enter ATAMS Extension. However, 74 subjects were included in ATAMS Extension and 1 subject could not enter due to the premature termination of the trial.
Groups:
- Atacicept 25 mg (With Loading): Subjects who received atacicept 25 milligram (mg) subcutaneously (SC) as loading dose twice weekly for first 4 weeks, followed by atacicept 25 mg SC for 32 weeks, in 28063 study were continued with atacicept 25 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
- Atacicept 75 mg (With Loading): Subjects who received atacicept 75 mg SC as loading dose twice weekly for first 4 weeks, followed by atacicept 75 mg SC for 32 weeks, in 28063 study were continued with atacicept 75 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
- Atacicept 150 mg (With Loading): Subjects who received atacicept 150 mg SC as loading dose twice weekly for first 4 weeks, followed by atacicept 150 mg SC for 32 weeks, in 28063 study were continued with atacicept 150 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
- Atacicept 150 mg (Without Loading): Subjects who received placebo SC twice weekly for first 4 weeks, followed by placebo SC for 32 weeks, in 28063 study were continued with atacicept 150 mg (without loading dose) SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
Period: Overall Study
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Started | 16 | 19 | 17 | 22
Completed | 0 | 0 | 0 | 0
Not Completed | 16 | 19 | 17 | 22
Not completed — Premature Termination | 16 | 15 | 14 | 21
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other | 0 | 2 | 0 | 0
Not completed — Randomised but not Treated | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized subjects.
Groups:
- Atacicept 25 mg (With Loading): Subjects who received atacicept 25 mg SC as loading dose twice weekly for first 4 weeks, followed by atacicept 25 mg SC for 32 weeks, in 28063 study were continued with atacicept 25 mg SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
- Total: Total of all reporting groups
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading) | Total
Number analyzed (Participants) | 16 | 19 | 17 | 22 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (8.4) | 36.8 (9.1) | 37.4 (11.2) | 34.4 (8.6) | 36.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 8 | 16 | 44
  Male | 8 | 7 | 9 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Injection Site Reactions, Infections, and Malignancies by Severity
Description: TEAEs were defined as AEs with a start date after or on the date of the first DB treatment injection in ATAMS Extension and that occurred anytime after treatment discontinuation, or up to the day before first Rebif® rescue medication injection in ATAMS Extension. A serious TEAE was an AE that resulted in any of the following: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE severity was graded as per Qualitative Toxicity Scale. Local injection site reactions (injection site: pain, redness, itching and swelling) throughout ATAMS Extension, starting after the first trial medication administration. If the subject experienced 1 or more of the above injection site symptoms, these were reported with the AE verbatim term "injection site reaction". For all randomized subjects, there was an option of rescue treatment with Rebif® for 1 year beginning with the first injection of Rebif®).
Time Frame: From the first dose of study drug administration up to Week 24
Population: Double-blind safety analysis set included all the subjects who received at least 1 dose of trial medication in the ATAMS extension study.
Measure: Number; unit: Subjects
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 17 | 15 | 22
Subjects
  Mild TEAEs | 5 | 8 | 8 | 13
  Moderate TEAEs | 2 | 4 | 6 | 4
  Severe TEAEs | 0 | 0 | 0 | 1
  Mild serious TEAEs | 0 | 0 | 0 | 0
  Moderate serious TEAEs | 0 | 1 | 0 | 0
  Severe serious TEAEs | 0 | 0 | 0 | 0
  Mild injection site reaction | 2 | 2 | 5 | 5
  Moderate injection site reaction | 0 | 0 | 0 | 2
  Severe injection site reaction | 0 | 0 | 0 | 0
  Mild infections | 1 | 2 | 4 | 6
  Moderate infections | 0 | 1 | 2 | 0
  Severe infections | 0 | 0 | 0 | 0
  Mild malignancies | 0 | 0 | 0 | 0
  Moderate malignancies | 1 | 0 | 0 | 0
  Severe malignancies | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure (systolic and diastolic) was measured after at least 3 minutes resting, with the subject in the seated position.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24 and 36
Population: Double-blind safety analysis set included all the subjects who received at least 1 dose of trial medication in the ATAMS extension study. Here 'n' signifies those subjects who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 17 | 15 | 22
millimeter of mercury (mmHg)
  SBP: Week 2 (n = 13, 16, 14, 20) | 2.6 (8.3) | -3.0 (9.5) | -1.2 (10.7) | -0.2 (9.8)
  SBP: Week 4 (n = 15, 14, 12, 21) | 2.1 (7.9) | -2.4 (13.7) | -5.1 (12.6) | -0.1 (9.9)
  SBP: Week 8 (n = 13, 11, 12, 16) | 0.8 (10.5) | -2.1 (12.0) | -1.1 (12.5) | 0.4 (11.0)
  SBP: Week 12 (n = 11, 12, 8, 16) | 3.0 (11.7) | -5.8 (15.3) | -3.4 (10.2) | -0.9 (11.3)
  SBP: Week 16 (n=7, 9, 6, 12) | 5.9 (13.4) | -9.0 (18.6) | -2.0 (12.2) | -2.3 (10.0)
  SBP: Week 20 (n=3, 7, 2, 6) | 2.0 (23.1) | -9.7 (14.8) | -0.5 (0.7) | 3.3 (6.0)
  SBP: Week 24 (n=2, 4, 1, 6) | 5.0 (7.1) | -5.0 (4.1) | 10.0 (NA) — Standard deviation is not evaluable as only 1 subject was evaluated for this parameter. | -5.3 (7.7)
  SBP: Week 36 (n=0, 1, 0, 0) | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available. | -18.0 (NA) — Standard deviation is not evaluable as only 1 subject was evaluated for this parameter. | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available. | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available.
  DBP: Week 2 (n=15, 13, 14, 21) | -2.1 (8.2) | -1.9 (8.4) | -3.6 (10.6) | 0.3 (8.6)
  DBP: Week 4 (n=15, 14, 12, 21) | -0.5 (9.0) | -0.4 (8.7) | -5.1 (9.2) | 0.1 (7.7)
  DBP: Week 8 (n=13, 11, 12, 16) | -2.8 (7.7) | -1.6 (8.7) | -5.9 (10.2) | 0.1 (11.0)
  DBP: Week 12 (n=11, 12, 8, 16) | -3.8 (11.1) | -4.8 (8.1) | -3.5 (9.9) | -2.4 (10.3)
  DBP: Week 16 (n=7, 9, 6, 12) | -1.6 (14.2) | -2.9 (9.0) | -2.3 (4.2) | -1.6 (7.7)
  DBP: Week 20 (n=3, 7, 2, 6) | -2.0 (17.1) | -4.4 (6.0) | 2.0 (4.2) | 3.7 (6.3)
  DBP: Week 24 (n=2, 4, 1, 6) | 0.0 (0.0) | -6.3 (2.5) | 0.0 (NA) — Standard deviation is not evaluable as only 1 subject was evaluated for this parameter. | -1.0 (9.8)
  DBP: Week 36 (n=0, 1, 0, 0) | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available. | -8.0 (NA) — Standard deviation is not evaluable as only 1 subject was evaluated for this parameter. | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available. | NA (NA) — The number of subjects evaluated was zero. Hence, data is not available.

3. Primary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24 and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 17 | 15 | 22
beats per minute (beats/min)
  Week 2 (n=15, 13, 14, 21) | -2.1 (5.1) | -3.5 (5.5) | -3.8 (10.4) | 3.6 (11.4)
  Week 4 (n=15, 14, 12, 21) | 0.6 (8.7) | -0.6 (9.2) | 0.7 (8.2) | 2.0 (8.0)
  Week 8 (n=13, 11, 12, 16) | -1.7 (9.2) | -3.4 (9.1) | 1.3 (8.7) | 4.4 (12.4)
  Week 12 (n=11, 12, 8, 16) | -0.5 (6.2) | 0.7 (9.5) | -1.5 (8.9) | 4.5 (9.5)
  Week 16 (n=7, 9, 6, 12) | 3.9 (4.7) | 1.1 (10.5) | -0.2 (4.8) | 3.8 (9.1)
  Week 20 (n=3, 7, 2, 6) | -0.3 (2.1) | 3.9 (8.3) | -5.0 (9.9) | 11.0 (8.8)
  Week 24 (n=2, 4, 1, 6) | 2.5 (0.7) | -5.3 (9.4) | -22.0 (NA) — Standard deviation is not applicable as only 1 subject was evaluable for this parameter | 9.0 (5.3)
  Week 36 (n=0, 1, 0, 0) | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available. | 7.0 (NA) — Standard deviation is not applicable as only 1 subject was evaluable for this parameter | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available. | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available.

4. Primary Outcome: Change From Baseline in Vital Signs: Temperature
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24 and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 17 | 15 | 22
Degree Celsius
  Week 2 (n=15, 13, 14, 21) | -0.09 (0.27) | 0.09 (0.27) | 0.03 (0.21) | -0.07 (0.36)
  Week 4 (n=15, 14, 12, 21) | -0.03 (0.24) | 0.05 (0.42) | 0.03 (0.24) | -0.12 (0.31)
  Week 8 (n=13, 11, 12, 16) | -0.03 (0.40) | 0.05 (0.10) | 0.03 (0.28) | -0.14 (0.25)
  Week 12 (n=11, 12, 8, 16) | 0.02 (0.19) | 0.08 (0.36) | 0.09 (0.57) | -0.15 (0.34)
  Week 16 (n=7, 9, 6, 12) | -0.10 (0.21) | 0.17 (0.35) | -0.05 (0.23) | 0.01 (0.42)
  Week 20 (n=3, 7, 2, 6) | -0.37 (0.35) | 0.16 (0.56) | -0.25 (0.07) | -0.08 (0.45)
  Week 24 (n=2, 4, 1, 6) | 0.05 (0.07) | 0.30 (0.59) | 0.00 (NA) — Standard deviation is not applicable as only 1 subject was evaluable for this parameter. | -0.07 (0.26)
  Week 36 (n=0, 1, 0, 0) | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available. | 0.70 (NA) — Standard deviation is not applicable as only 1 subject was evaluable for this parameter. | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available. | NA (NA) — The number of subjects evaluable was zero. Hence, data is not available.

5. Primary Outcome: Change From Baseline in Electrocardiogram (ECGs)
Time Frame: Baseline, Week 12 and 36
Population: No summary tables were prepared for ECG parameters, and ECG data were not formally analyzed. However, a qualitative assessment of ECG morphology and rhythm was made by the Investigator and recorded in the electronic case report form (eCRF). ECG abnormalities considered significant by the investigator were reported as AEs.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Worsened Post Baseline Shift in Immunoglobulin A (IgA), IgG and IgM Levels
Description: Number of subjects with shifts from normal Grade (Grade 0) at Baseline to worse value at post-baseline (Grade 1 to Grade 4) according to the following criteria: IgA Grade 0: greater than or equal to (>=) lower limit normal (LLN) 0.7 gram per liter (g/L); Grade 1: less than (<) LLN - 0.5 g/L, Grade 2: <0.5g/L -0.3 g/L, Grade 3: <0.3 g/L -0.1 g/L, Grade 4: < 0.1 g/L; IgG Grade 0: >= LLN (7 g/L), Grade 1: < LLN - 5 g/L, Grade 2: <5g/L -4 g/L, Grade 3: <4 g/L -3 g/L and Grade 4: < 3 g/L; IgM Grade 0: >= LLN (0.4 g/L), Grade 1: < LLN - 0.3 g/L, Grade 2: <0.3 g/L -0.2 g/L, Grade 3: <0.2 g/L -0.1 g/L, and Grade 4: < 0.1 g/L are presented in this outcome measure.
Time Frame: Baseline up to Week 36
Population: Intent-to-treat (ITT) population included all randomized subjects.
Measure: Number; unit: Subjects
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 19 | 17 | 22
Subjects
  IgA | 1 | 3 | 10 | 9
  IgG | 4 | 8 | 12 | 5
  IgM | 7 | 6 | 14 | 7

7. Secondary Outcome: Number of Subjects With Clinical Attacks/Relapses
Description: A clinical attack/relapse was defined as the fulfillment of all the following criteria:
  1. Neurological abnormality, either newly appearing or re-appearing, with abnormality specified by both i) neurological abnormality separated by at least 30 days from onset of a preceding clinical event, and ii) neurological abnormality lasting for at least 24 hours.
  2. Absence of fever or known infection (fever with temperature (axillary, orally, or intra-auriculary) > 37.5°C/99.5 °Fahrenheit).
  3. Objective neurological impairment, correlating with the subject's reported symptoms, defined as either i) increase in at least 1 of the functional systems of the Expanded Disability Status Scale (EDSS), or ii) increase of the total EDSS score. EDSS overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Baseline up to Week 24
Population: Intent-to-treat (ITT) population included all randomized subjects.
Measure: Number; unit: Subjects
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 19 | 17 | 22
Subjects
  No Relapse | 16 | 16 | 15 | 21
  1 Relapse | 0 | 3 | 2 | 1
  2 Relapse | 0 | 0 | 0 | 0
  3 Relapse | 0 | 0 | 0 | 0
  Greater than or equal to (>=) 4 Relapse | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Scores at Week 12
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with multiple sclerosis (MS). It assesses the 8 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder, cerebral and other) as well as ambulation. EDSS overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) population included all randomized subjects. "N" signifies (total number of subjects analyzed) the number of evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 11 | 13 | 10 | 16
Units on a scale | 0.09 (0.58) | 0.04 (0.97) | 0.50 (0.85) | -0.06 (0.75)

9. Secondary Outcome: Change in Multiple Sclerosis Functional Composite (MSFC) Score at Week 12
Description: The MSFC is a multidimensional clinical outcome measure which consists of three sub-tests; Timed 25-Foot Walk, 9-Hole Peg Test and Paced Auditory Serial Addition Test-3(PASAT-3). The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The 9-Hole Peg Test is a quantitative measure of upper extremity (arm and hand) function. The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Standardized results (Z-scores) of these sub-tests and the overall MSFC Z-score as an average of these three Z-scores was calculated. Higher Z-scores reflect better neurological function and a positive change from baseline indicates improvement. An increase in score indicates an improvement (range -3 to +3).
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all randomized subjects. "N" signifies number of evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 11 | 13 | 9 | 16
z-score | 0.21 (0.40) | 0.04 (0.47) | -0.01 (0.24) | 0.07 (0.34)

10. Secondary Outcome: Magnetic Resonance Imaging (MRI) Parameters: Number of T1 Gadolinium (Gd)-Enhancing Lesions Per Subject
Time Frame: Baseline, Week 12 and 24
Population: Intent-to-treat (ITT) population included all randomized subjects. "n" signifies the number of evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of lesions per subject
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 19 | 17 | 22
Number of lesions per subject
  Baseline (n=16, 19, 17, 22) | 1.1 (2.2) | 2.3 (5.0) | 0.8 (1.4) | 0.9 (1.4)
  Week 12 (n=11, 11, 7, 15) | 0.27 (0.47) | 0.64 (1.29) | 1.00 (1.15) | 2.27 (7.16)
  Week 24 (n=2, 3, 1, 6) | 0.00 (0.00) | 2.00 (2.00) | 0.00 (0.00) | 0.83 (0.75)

11. Secondary Outcome: Magnetic Resonance Imaging (MRI) Parameters: Volume of T2 Lesions (New or Enlarging T2 Lesions) Per Subject
Time Frame: Baseline, Week 12 and Week 24
Measure: Mean (Standard Deviation); unit: Cubic millimeter
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 16 | 19 | 17 | 22
Cubic millimeter
  Baseline (n=16, 19, 17, 22) | 4792.76 (3152.56) | 8196.59 (8888.74) | 6158.04 (7945.59) | 5868.84 (7170.81)
  Week 12 (n=11, 11, 7, 15) | 5604.42 (5154.52) | 7634.89 (6340.19) | 4934.03 (4802.98) | 5365.63 (7445.87)
  Week 24 (n=2, 3, 1, 6) | 1699.60 (586.76) | 6814.60 (6643.00) | 1931.40 (0.00) | 5541.80 (5614.73)

12. Secondary Outcome: Concentrations of Free and Total Atacicept
Time Frame: Baseline and Week 12
Population: This outcome measure was not assessed due to lack of a valid assay during the usable time period of the samples.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Free B-Lymphocyte Stimulator (BLyS) and Free A Proliferation-Inducing Ligand (APRIL) Serum Concentrations.
Description: Levels of free APRIL and free BLyS: Free APRIL serum samples were to be analyzed by using a validated enzyme-linked immunosorbent assay (ELISA) with limits of detection of 0.3125 nanogram per milliliter (ng/mL) for free APRIL and free BlyS serum samples were analysed using a validated ELISA with limits of detection of 1.56 ng/mL.
Time Frame: Baseline, Week 12 and 36
Population: This outcome measure was not assessed due to lack of a valid assay for measuring BLyS and APRIL.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Pharmacogenetics/Pharmacogenomics Analysis
Description: Gene expression profiling and gene polymorphism identification were to be used to identify putative markers for response to treatment.
  * Genome-wide gene polymorphism characterization by genome-wide scan.
  * Targeted gene polymorphism identification of B-Lymphocyte Stimulator (BLyS) , APRIL, (receptor for B cell activating factor of the tumor necrosis factor [TNF] family) BAFF-R, (Transmembrane Activator) TACI and (B Cell Maturation Antigen) BCMA and HLA-DRB1 by direct genotyping or sequencing .
Time Frame: Day 1 and Week 36
Population: Genetic/genomic analysis was not performed as the trial was terminated early.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Subjects With Positive Neutralizing Antibody (NAb)
Time Frame: Baseline, Week 12 and 36
Population: Appropriate method/test was not established to identify the positive neutralizing antibodies for atacicept. Hence, this outcome measure was not assessed.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to Week 24
Description: AEs were collected for Double-blind safety analysis set which included all the subjects who received at least 1 dose of trial medication in the ATAMS extension study.
Groups:
- Atacicept 150 mg (Without Loading): Subjects who received placebo SC as loading dose twice weekly for first 4 weeks, followed by placebo SC for 32 weeks, in 28063 study were continued with atacicept 150 mg (without loading dose) SC once weekly up to 5 years or up to early termination of treatment or early termination of the study.
Arm/Group | Atacicept 25 mg (With Loading) | Atacicept 75 mg (With Loading) | Atacicept 150 mg (With Loading) | Atacicept 150 mg (Without Loading)
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/17 | 0/15 | 0/22
Other Adverse Events (participants affected / at risk) | 6/16 | 9/17 | 8/15 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 25 mg (With Loading) (N=16) | Atacicept 75 mg (With Loading) (N=17) | Atacicept 150 mg (With Loading) (N=15) | Atacicept 150 mg (Without Loading) (N=22)
Peripheral Edema (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 25 mg (With Loading) (N=16) | Atacicept 75 mg (With Loading) (N=17) | Atacicept 150 mg (With Loading) (N=15) | Atacicept 150 mg (Without Loading) (N=22)
Injection site reaction (General disorders) | 2 | 2 | 5 | 7
Fatigue (General disorders) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 1
Bilirubin urine (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0
Creatinine renal clearance increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Tic (Psychiatric disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Sponsor voluntarily decided to terminate this trial after observing increased MS disease activity in trial 28063 ATAMS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study as a whole will be published prior to any individual investigator publications. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.